CLINICAL TRIAL: NCT01512576
Title: Does Acupuncture Activate Endogenous Pain Inhibition in Chronic Whiplash Associated Disorders? A Randomized Cross-over Trial
Brief Title: Does Acupuncture Activate Endogenous Pain Inhibition in Chronic Whiplash?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Jo Nijs, Associate professor, Vrije Universiteit Brussel
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AcuWAD
Record Dates: First submitted 2012-01-11; First posted 2012-01-19 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: Whiplash
Keywords: whiplash; chronic pain; sensitization; treatment; acupuncture; relaxation
MeSH Terms: conditions — Whiplash Injuries; Chronic Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- acupuncture (Experimental): All patients were treated at the basic points bilaterally situated in the local region (neck), distal region (low back, arms and legs) and ear. In addition, acupuncture treatment was performed according to the rules of traditional Chinese medicine and was semi-standardized. This means that the therapist was allowed to choose from a list of the following acupuncture points: GV14, Huatuojiaji C1-C7, GB20, SI11, GB21, TE15, SI14, BL17, MT10, SI3, BL64, TE5, GB41, Zero point, Jerome point, C0. The combination of acupuncture points were chosen individually, according to the patients' self-reported symptoms. In order to obtain the required information, patients had to fill out a Margolis pain diagram, and the acupuncturist questioned the patient and performed a tongue- and pulse diagnosis.
  Interventions: Other: acupuncture
- relaxation (Active Comparator): For the relaxation treatment the method of guided imagery is applied. Guided imagery is a system of visualization. During guided imagery relaxation, the patient's state of consciousness is similar to one which occurs in meditative status. Patients are instructed to listen to a CD with relaxation music (Arcade TV-CD Ad Vissesr's Brainsessions, track 3). Patients will sit in an identical position like during the acupuncture treatment (i.e. on a relaxation chair) and listened to the audio CD by headphone.
  Interventions: Behavioral: relaxation

INTERVENTIONS:
Other: acupuncture — one 30-minute treatment session using sterile 1-time-use needles (Euro-acupuncture needles) were used, but the therapist was allowed to chose the needle length and diameter
  Other Names: complex somatosensory stimulation
  Arms: acupuncture
Behavioral: relaxation — 1 treatment session of 30 minutes
  Other Names: visualization
  Arms: relaxation

SUMMARY:
This physiological study examines whether acupuncture exerts short-term effects of analgesic mechanisms in patients with chronic whiplash pain. More specifically, it is examined whether acupuncture activates brain-orchestrated pain inhibitory action.

DETAILED DESCRIPTION:
Many patients with chronic pain, including those with chronic whiplash-associated disorders (WAD), show features of central sensitization (CS), a process characterized by generalized hypersensitivity of the somatosensory system. it would be worthwhile identifying treatments able of activating the dysfunctional endogenous pain inhibition in patients with CS and chronic WAD.

Acupuncture is a treatment method widely used for patients with chronic pain, including those with chronic WAD. The effectiveness of acupuncture for the treatment of chronic (neck) pain is supported by several randomized controlled clinical trials, systematic reviews including meta-analyses. However, the effect-sizes are rather small and only short-term effects have been shown consistently.

A randomized cross-over trial comparing acupuncture with relaxation is conducted in order to examine whether acupuncture vs. relaxation for patients with chronic WAD results in:

1. Immediate activation of endogenous pain inhibition (i.e. conditioned pain modulation);
2. Concomitant pain relief;
3. And reduced disability level. Further it is examined whether acupuncture vs. relaxation results in different autonomic nervous system responses.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of chronic WAD grade 1 to 3 according to the criteria as defined by the Quebec Task Force classification
* chronic neck pain and WAD persisting for at least 3 months
* age between 18 and 65 years

Exclusion Criteria:

* classified as WAD grade 4 (neck complaints including fracture or dislocation, or injury to the spinal cord)
* pregnant
* initiated a new conventional therapy during the study period
* taking analgesic drugs 48 hours before testing and/or nicotine, alcohol and caffeine 24 hours before testing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
the change in Conditioned pain modulation | measured prior to (week 1 and week 2) and immediately following (week1 and week 2) each treatment session
  For assessing CPM, the method examining the influence of the Diffuse Noxious Inhibitory Control system (or spatial summation) on temporal summation (TS) was applied. The experimental pain assessments before and after each treatment were carried out by the same assessor.

SECONDARY OUTCOMES:
the change in Neck Disability Index (NDI) | measured prior to (week 1 and 2) and immediately following (week 1 and 2) each treatment session
  The Neck Disability Index (NDI) was developed in 1991 as a modification of the Oswestry Back Pain Index and was the first instrument designed to assess self-rated disability in patients with neck pain. The NDI is scored from 0 (good function) to 50 (poor function) and when multiplied by two the percentage of disability can be obtained. The NDI is a valid and reliable instrument, sensitive to measure changes within a population of patient with neck pain.
the change in autonomic activity | week 1 and 2 : measured continuously in real time during CPM and during both treatment sessions
  For measuring autonomic activity, the Nexus 10 device (Mind Media, the Netherlands) will be used. Skin conductance, body temperature, heart rate, blood volume pressure and heart rate variability will be measured continuously in real time during CPM and during both treatment sessions. Electrodes will be placed on the left hand in all patients.
the change in scores obtained from the Whiplash Associated Disorders Symptom List | measured prior to (week 1 and 2) and immediately following (week 1 and 2) each treatment session
  The Whiplash Associated Disorders Symptom List is a self-reported measure for assessing symptom severity in WAD patients. The questionnaire is composed of the most frequently reported WAD symptoms in the literature and some autonomic symptoms. Every symptom is presented by a visual analogue scale (VAS) (100 mm), a method that is known for its validity and reliability.

CONTACTS AND LOCATIONS:
Overall Officials: Jo Nijs, PhD, Principal Investigator — Vrije Universiteit Brussel
Locations (1):
- Vrije Universiteit Brussel, Brussels, Belgium

REFERENCES:
- [Background] Nijs J, Meeus M, Van Oosterwijck J, Roussel N, De Kooning M, Ickmans K, Matic M. Treatment of central sensitization in patients with 'unexplained' chronic pain: what options do we have? Expert Opin Pharmacother. 2011 May;12(7):1087-98. doi: 10.1517/14656566.2011.547475. Epub 2011 Jan 22. PMID 21254866
- [Background] Nijs J, Van Oosterwijck J, De Hertogh W. Rehabilitation of chronic whiplash: treatment of cervical dysfunctions or chronic pain syndrome? Clin Rheumatol. 2009 Mar;28(3):243-51. doi: 10.1007/s10067-008-1083-x. Epub 2009 Jan 22. PMID 19160000
- [Background] Nijs J, Inghelbrecht E, Daenen L, Hachimi-Idrissi S, Hens L, Willems B, Roussel N, Cras P, Wouters K, Bernheim J. Recruitment bias in chronic pain research: whiplash as a model. Clin Rheumatol. 2011 Nov;30(11):1481-9. doi: 10.1007/s10067-011-1829-8. Epub 2011 Aug 19. PMID 21853277